CLINICAL TRIAL: NCT02114879
Title: Enhanced Medical Rehabilitation in Older Adults
Acronym: EMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 MH099011A1; 5R01MH099011-02 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-15 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Disabling Medical Events; Disabled; Depression
Keywords: Physical Therapy; Occupational Therapy; Rehabilitation; Older adults; Depression; Physical Functioning
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Rehabilitation (Active Comparator)
  Interventions: Behavioral: Standard of Care Rehabilitation
- Enhanced Medical Rehabilitation (Experimental)
  Interventions: Behavioral: Enhanced Medical Rehabilitation

INTERVENTIONS:
Behavioral: Enhanced Medical Rehabilitation — Daily PT/OT provided by therapists trained in Enhanced Medical Rehabilitation. This training focuses on improved communication, patient engagement, and intensity.
  Arms: Enhanced Medical Rehabilitation
Behavioral: Standard of Care Rehabilitation — Daily PT/OT provided by therapists not trained in the treatment intervention.
  Arms: Standard of Care Rehabilitation

SUMMARY:
The purpose of this study is to provide evidence that Enhanced Medical Rehabilitation is an effective treatment for older adults after disabling medical events.

DETAILED DESCRIPTION:
The intervention involves physical and occupational therapy for patients who have been admitted to a skilled nursing facility for therapy following a disabling medical event.

Participants in this study will be randomly assigned to receive either Enhanced or standard of care therapy, meaning they will either receive their PT (Physical Therapy)& OT(Occupational Therapy) from therapists who have been specially trained in the study intervention or from therapists with normal training. Participants will be assessed at baseline, 30, 60, and 90 days after baseline, and at the date of their discharge from the skilled nursing facility.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* Admitted to a skilled nursing facility for post-acute care from PT and OT for 2 weeks or more.

Exclusion Criteria:

* Language, visual or hearing barriers to participation
* Medical illness preventing study participation or accurate data collection
* Moderate-severe dementia (demonstrated by chart diagnosis and/or short blessed score greater than 13)
* Progressive neurological condition such that recovery of function is not feasible
* Patient did not have the ability to walk prior to hospitalization (e.g. paraplegic)
* Schizophrenia or other chronic or current psychotic disorder.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Barnes-Jewish Extended Care, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Alexian Brothers Sherbrooke Village, St Louis, Missouri

REFERENCES:
- [Background] Bland MD, Birkenmeier RL, Barco P, Lenard E, Lang CE, Lenze EJ. Enhanced Medical Rehabilitation: Effectiveness of a clinical training model. NeuroRehabilitation. 2016 Oct 14;39(4):481-498. doi: 10.3233/NRE-161380. PMID 27689608
- [Derived] Ercal B, Rodebaugh TL, Bland MD, Barco P, Lenard E, Lang CE, Miller JP, Yingling M, Lenze EJ. Executive Function Moderates Functional Outcomes of Engagement Strategies During Rehabilitation in Older Adults. Am J Phys Med Rehabil. 2021 Jul 1;100(7):635-642. doi: 10.1097/PHM.0000000000001739. PMID 34131093
- [Derived] Lenze EJ, Lenard E, Bland M, Barco P, Miller JP, Yingling M, Lang CE, Morrow-Howell N, Baum CM, Binder EF, Rodebaugh TL. Effect of Enhanced Medical Rehabilitation on Functional Recovery in Older Adults Receiving Skilled Nursing Care After Acute Rehabilitation: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jul 3;2(7):e198199. doi: 10.1001/jamanetworkopen.2019.8199. PMID 31365113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 skilled nursing facilities in the St. Louis, Missouri metropolitan area from July 29, 2014 through March 22, 2018.
Period: Overall Study
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Started | 115 | 114
Completed | 96 | 90
Not Completed | 19 | 24
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Death | 6 | 11
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation | Total
Number analyzed (Participants) | 115 | 114 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (7.7) | 79.5 (8.2) | 79.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 114 | 114 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 25 | 51
  White | 89 | 88 | 177
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Impairment Type [Count of Participants; unit: Participants] — Participants' medical conditions were rated by organ system using the Cumulative Illness Rating Scale for Geriatrics (CIRS-G). Participants with extremely severe impairment (CIRSG item score of 4) are tabulated below. Some participants had extremely severe impairment in more than one category.
  Participants
    Musculoskeletal/Integument | 44 | 36 | 80
    Heart | 29 | 31 | 60
    Respiratory | 18 | 25 | 43
    Renal | 7 | 7 | 14
    Neurologic | 5 | 5 | 10
    Other/Unknown | 22 | 19 | 41
MADRS Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a measurement of depressive symptom severity. Scores can range from 0-60 with higher scores indicating more depressive symptoms.
  units on a scale | 8.4 (8.0) | 8.8 (7.6) | 8.6 (7.8)
Short Blessed Test Score [Mean (Standard Deviation); unit: units on a scale] — The Short Blessed Test is a measure of cognitive impairment. It is a brief assessment of orientation, registration, and attention. Scores range from 0-28. Higher scores indicate worse impairment, with scores of 5-9 consistent with mild cognitive impairment and scores of at least 10 consistent with dementia.
  units on a scale | 3.8 (3.2) | 4.4 (3.6) | 4.1 (3.4)
Barthel Index Total Score (Premorbid) [Mean (Standard Deviation); unit: units on a scale] — The Barthel Index is an instrument that measures a person's ability to perform 10 basic activities of daily living or mobility items, with a scale range between 0 and 100 (higher scores indicate better function).
  units on a scale | 95.1 (9.0) | 96.1 (6.9) | 95.6 (8.1)
Barthel Index Total Score (Admission) [Mean (Standard Deviation); unit: units on a scale] — The Barthel Index is an instrument that measures a person's ability to perform 10 basic activities of daily living or mobility items, with a scale range between 0 and 100 (higher scores indicate better function).
  units on a scale | 34.7 (12.8) | 32.3 (13.1) | 33.5 (13.0)
CIRS-G Score [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) is used to quantify chronic illness burden from the medical records. Higher scores indicate greater burden.
  units on a scale | 17.1 (5.4) | 16.8 (5.0) | 16.9 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Barthel Index Score
Description: Barthel Index scores range from 0 to 100, with higher scores indicating greater levels of function.
Time Frame: Baseline and Discharge, an average of 24 days.
Population: One Standard of Care participant did not have a baseline Barthel completed. Otherwise, all other 228 participants were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 114 | 114
score on a scale | 28.48 (1.68) | 34.92 (1.66)
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; This Primary analysis used a marginal model with time (baseline and discharge), condition (EMR vs SOC), and time x condition as fixed effects, with an unstructured covariance structure specified, based on Bayesian information criteria (BIC); Test type: Superiority; p = 0.007, Marginal Model — The p-value refers to the time by group interaction. The a priori threshold for statistical significance in this planned primary test was p<0.05

2. Secondary Outcome: Gait Speed (Determined by 4 or 10 Meter Walk Test)
Description: Meters walked per second.
Time Frame: Discharge, an average of 24 days after baseline.
Population: All participants with a gait speed at discharge were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: meters per second
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 94 | 105
meters per second | 0.45 [0.13 to 0.63] | 0.35 [0.05 to 0.52]
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Distance Ambulated in 6-Minute Walk Test
Description: Feet walked during 6 minute interval.
Time Frame: Discharge, an average of 24 days after baseline.
Population: All participants able to perform a 6-minute walk at discharge were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: feet
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 93 | 104
feet | 210 [53.00 to 354.50] | 170 [41.75 to 364.50]
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Self-reported Barthel Index
Description: Barthel Index scores range from 0 to 100, with higher scores indicating greater levels of function. Conducted as a self-report at timepoints where patient was not in an institutional setting.
Time Frame: 30, 60, and 90 Days Post Admission to the SNF
Population: Any participant with data at either 30 days, 60 days, 90 days, or at discharge were included in the analyses.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 114 | 114
score on a scale
  Day 30 | 78.95 (2.08) | 78.79 (2.08)
  Day 60 | 85.01 (1.94) | 84.27 (1.99)
  Day 90 | 84.67 (2.16) | 83.65 (2.20)
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.96, Mixed Models Analysis — The p-value refers to the time by group interaction. The statistical significance in this test was p<0.05

5. Secondary Outcome: Discharge Disposition
Description: Number of participants discharged from skilled nursing facility to home
Time Frame: Discharge, an average of 24 days after baseline.
Population: Any participant with a discharge disposition of either 'to home' or 'to institution' were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 110 | 110
Participants | 89 | 94
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; Test type: Superiority; p = 0.37, Chi-squared — The p-value is calculated from a 2x2 Contingency Table consisting of rows that represent Discharged Home Vs Discharged to Institution and columns that represent the EMR and SOC groups

6. Secondary Outcome: Rehospitalizations
Description: Assesses whether the participant was readmitted to the hospital.
Time Frame: Days 30, 60, and 90 post admission to a SNF as well as at Discharge
Population: Any participant with at least one re-hospitalization at day 30, day 60, day 90 or at discharge was included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
Number analyzed (Participants) | 110 | 111
Participants | 43 | 42
Statistical Analysis 1: Comparison: Standard of Care Rehabilitation vs Enhanced Medical Rehabilitation; Test type: Superiority; p = 0.85, Chi-squared — The p-value is calculated from a 2x2 Contingency Table consisting of rows that represent Yes/No Rehospitalization and columns that represent the EMR and SOC groups

ADVERSE EVENTS:
Time Frame: 90 days
Description: All cause mortality was tracked for 90 days.
Arm/Group | Standard of Care Rehabilitation | Enhanced Medical Rehabilitation
All-Cause Mortality (participants affected / at risk) | 6/115 | 11/114
Serious Adverse Events (participants affected / at risk) | 6/115 | 11/114
Other Adverse Events (participants affected / at risk) | 0/115 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Rehabilitation (N=115) | Enhanced Medical Rehabilitation (N=114)
all cause mortality (General disorders) | 6 (6) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT02114879/SAP_000.pdf
  • Study Protocol (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02114879/Prot_001.pdf